CLINICAL TRIAL: NCT01690767
Title: A Randomized Blinded Controlled Trial of 2% Lidocaine Gel Compared to Standard of Care in Children Undergoing Urethral Catheterization
Brief Title: A Study to Assess the Ability of 2% Lidocaine Gel to Reduce the Discomfort of Urethral Catheterization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Naveen Poonai, Attending Physician, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17770
Record Dates: First submitted 2011-02-15; First posted 2012-09-24 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Urinary Tract Infection
Keywords: Urethral catheterization; Lidocaine
MeSH Terms: conditions — Urinary Tract Infections | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical and intraurethral 2% lidocaine (Experimental): 2% lidocaine gel will be applied for 5 minutes to the external urethral opening. This will be followed immediately by 2% lidocaine gel administration into the urethra using a 24 gauge angiocath for 5 minutes prior to catheterization for urine specimen collection. Children < 7 kg and > 7 kg will receive 1 cc and 1.5 cc, respectively.
  Interventions: Drug: 2% lidocaine gel
- Standard of care (Active Comparator): According to standard nursing practice, the urethra will be catheterized without anaesthetic gel but using lubricant gel only. Intervention is Health Care Lubricating Jelly.
  Interventions: Drug: Health Care Lubricating Jelly

INTERVENTIONS:
Drug: 2% lidocaine gel — Children < 7 kg and > 7 kg will receive 1 cc and 1.5 cc of 2% lidocaine gel, respectively
  Other Names: Lidocaine
  Arms: Topical and intraurethral 2% lidocaine
Drug: Health Care Lubricating Jelly — Non-medicinal lubrication gel
  Other Names: Muco
  Arms: Standard of care

SUMMARY:
Children 0-24 months of age requiring a urethral catheterization for urine collection will be randomized to receive either topical and intraurethral 2% lidocaine or standard of care to assess for the effectiveness of the former in minimizing pain during urethral catheterization. It is hypothesized that administration of 2% lidocaine gel both topically and intraurethrally will confer a greater degree of pain reduction compared to standard of care.

DETAILED DESCRIPTION:
An estimated 10% of children 0-24 months of age that present to the emergency department (ED) with fever and/or vomiting have a urinary tract infection (UTI). An accurate diagnosis of a UTI ensures timely and appropriate treatment given to reduce the risk of renal scarring, which is the greatest in this age group. To ensure diagnostic accuracy, urethral catheterization is the preferred method to obtain a urine sample from a young child. In contrast to adults, most children do not receive local analgesia for urethral catheterization; despite growing recognition that children experience avoidable pain and discomfort during invasive procedures.

Following informed consent, participants will be randomized by block randomization in a concealed fashion to receive either topical and intraurethral 2% lidocaine or standard of care using a computerized random number generator. The research nurse will access a sequentially numbered, opaque sealed envelope that will contain the participant's group assignment. No adjunctive analgesic methods will be used. A research pharmacist will prepare 2% lidocaine gel in a 3 cc syringe attached to a 24 gauge angiocath. Children < 7 kg and > 7 kg will receive 1 cc and 1.5 cc, respectively (2).

The entire procedure will be videotaped and participants pain will be scored using a brow bulging score and visual analogue scale by independent, blinded raters.

ELIGIBILITY:
Inclusion Criteria:

* children 0-24 months of age presenting to the emergency department requiring a urethral catheterization to obtain a urine specimen

Exclusion Criteria:

* unstable
* external genitourinary anomalies
* lidocaine allergy and
* previous catheterization within 24 hours

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Brow Bulging Score | 30 seconds post intervention compared to baseline
  The presence of brow bulging will be scored in 2-second intervals for the first 30 seconds for each of the six phases. The percentage of time that brow bulging is observed will then be calculated for each phase.

SECONDARY OUTCOMES:
Facial grimacing score | 30 seconds post intervention compared to placebo
  The presence of brow bulging, nasolabial furrowing and eyes squeezing shut will be scored in 2-second intervals for the first 30 seconds for each of the six phases. The percentage of time that all three of these features is observed will then be calculated for each phase.

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Poonai, MD, FRCPC, Principal Investigator — Western University, Canada
Locations (1):
- Children's Hospital, London Health Sciences Center, London, Ontario, Canada

REFERENCES:
- [Derived] Poonai N, Li J, Langford C, Lepore N, Taddio A, Gerges S, Stitt L, Teefy J, Manji K, Castelo M, Rieder M, Qui T, Matsui D, Ali S. Intraurethral Lidocaine for Urethral Catheterization in Children: A Randomized Controlled Trial. Pediatrics. 2015 Oct;136(4):e879-86. doi: 10.1542/peds.2015-1852. PMID 26416942